CLINICAL TRIAL: NCT05635227
Title: Dexamethasone, Olanzapine, Flow-targeted Versus Pressure-targeted Hemodynamic Management, and Low Tidal Volume Ventilation in Patients Undergoing On-pump Cardiac Surgery - a Multifactorial Design Randomized Trial
Brief Title: Dexamethasone, Olanzapine, Hemodynamics, and Ventilation in Cardiac Surgery
Acronym: GLORIOUS-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sebastian Wiberg, Principal Investigator, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-HJEPharma-002
Record Dates: First submitted 2022-11-13; First posted 2022-12-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease; Aortic Valve Disease
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease | interventions — dexamethasone 21-phosphate; Sodium Chloride; Olanzapine

STUDY DESIGN:
Intervention Model Description: The trial assumes a priori that any effect of each of the four interventions are independent from any effect of another intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The dexamethasone intervention will be carried out by the nurse anesthetist and the perfusionist, and accordingly will be un-blinded. The perfusionists and the nurse anaesthetist will not be involved in any postoperative clinical care, outcome evaluation, or data analyses. The participant, trial staff, and all clinical personnel with the exception of the nurse anaesthetist and perfusionist will be blinded.
  The olanzapine intervention will be blinded for all; including the participant, trial staff, and all clinical personnel.
  The hemodynamic and ventilatory strategy interventions will be unblinded for the staff in the operating theatre (OR). The interventions will be blinded for the participants, trial staff and clinical personnel outside the OR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Dexamethasone (Experimental): The dexamethasone kit will contain 20 mg of dexamethasonphosfat (Dexavit®,Vital Pharma Nordic), 4mg/mL, i.e. 5 mL, which corresponds to 16.67 mg of dexamethasone. Dexamethasone will be administered as an intravenous bolus infusion over 2 minutes after induction of anaesthesia.
  Interventions: Drug: Dexamethasone phosphate
- Placebo (for Dexamethasone) (Placebo Comparator): The placebo kit will contain 5 mL of isotonic (0.9%) normal saline. Placebo will be administered as an intravenous bolus infusion over 2 minutes after induction of anaesthesia.
  Interventions: Drug: Isotonic sodium chloride (0.9%)
- Olanzapine (Experimental): The olanzapine kit will consist of two capsules each containing two 2.5 mg tablets of olanzapine (Olanzapine Stada®, STADA Nordic); i.e. total dose 10mg. The capsules will be delivered to the patient with instruction to take the capsule orally along with other standardized pre-procedure medicine. Patient intake will be recorded.
  Interventions: Drug: Olanzapine 10 MG
- Placebo (for Olanzapine) (Placebo Comparator): The placebo kit will consist of two placebo capsules identical to the capsules containing the olanzapine tablet. The capsules will be delivered to the patient with instruction to take the capsule orally along with other standardized pre-procedure medicine. Patient intake will be recorded.
  Interventions: Drug: Placebo capsule
- Flow-targeted hemodynamic management (Experimental): In the 'flow group', an arterial oxygen delivery (DO2) above 274 mL/min/m2 BSA AND a central venous oxygen saturation (ScvO2) above 70% will be targeted. CPB pump flow will be initiated at a flow rate of 2.4 L/min/m2. If DO2 or ScvO2 are below target, CPB pump flow will be gradually increased until targets are reached up to a maximum CPB pump flow of 3.2 L/min/m2. If DO2 or ScvO2 are below targets despite a maximum CPB pump flow, PaO2 will be gradually increased from an initial target of 15-20 kPa to a maximum of 40 kPa. A haematocrit level equal to or above 21% will be targeted, however, if DO2 or ScvO2 are below target despite a CPB pump flow of 3.2 L/min/m2, the haematocrit target level will be increased to equal to or above 25%. A MAP down to 35 mmHg will be tolerated throughout. The MAP target will be achieved by administration of boluses of phenylephrine up to a total of 2.0 mg, which can be followed by a continuous infusion of norepinephrine up to 0.6 μg per kg per min.
  Interventions: Procedure: Flow-targeted hemodynamic management
- Pressure-targeted hemodynamic management (Active Comparator): In the 'pressure group' a MAP between 70 to 80 mmHg will be targeted. The assigned MAP target will be achieved by administration of boluses of phenylephrine up to a total of 2.0 mg, which can be followed by a continuous infusion of norepinephrine up to 0.6 μg per kg per min. CPB pump flow will be fixed at a flow rate of 2.4 L per minute per square meter body surface area. A haematocrit level equal to or above 21% will be targeted throughout. A PaO2 of 15-20 kPa will be targeted throughout.
  Interventions: Procedure: Pressure-targeted hemodynamic management
- Low tidal-volume ventilation (Experimental): During initiation of CPB, the 'ventilation' group will receive a tidal volume at 3ml/kg and a set PEEP of 3 cm H2O. The respiratory frequency (RF) will be set at 10, and the inspiratory: expiratory (I:E) ratio will be set to 5:1. Peak pressures (Pmax) will be limited to < 25 cm H2O. FiO2 will be set at 50%. The ventilation strategy will be maintained during CPB.
  Any recruitment manoeuvres will be initiated solely at the discretion of the attending anaesthesiologist, and only if the patient's oxygen saturation drops below 88%. All recruitment manoeuvres will be completed by increasing the inspiratory pressure to 20 cmH2O for 10 seconds. The manoeuvre will be repeated three times.
  Interventions: Procedure: Low tidal-volume ventilation
- No ventilation (Active Comparator): The 'no-ventilation' group will receive no ventilation or PEEP. The ventilation strategy will be maintained during CPB.
  Any recruitment manoeuvres will be initiated solely at the discretion of the attending anaesthesiologist, and only if the patient's oxygen saturation drops below 88%. All recruitment manoeuvres will be completed by increasing the inspiratory pressure to 20 cmH2O for 10 seconds. The manoeuvre will be repeated three times.
  Interventions: Procedure: No ventilation

INTERVENTIONS:
Drug: Dexamethasone phosphate — See description of arms
  Arms: Dexamethasone
Drug: Isotonic sodium chloride (0.9%) — See description of arms
  Arms: Placebo (for Dexamethasone)
Drug: Olanzapine 10 MG — Olanzapine tablet pre-hidden in capsule identical to the placebo tablet
  Arms: Olanzapine
Drug: Placebo capsule — capsule identical to capsule containing olanzapine
  Arms: Placebo (for Olanzapine)
Procedure: Flow-targeted hemodynamic management — See description of arms
  Arms: Flow-targeted hemodynamic management
Procedure: Pressure-targeted hemodynamic management — See description of arms
  Arms: Pressure-targeted hemodynamic management
Procedure: Low tidal-volume ventilation — See description of arms
  Arms: Low tidal-volume ventilation
Procedure: No ventilation — See description of arms
  Arms: No ventilation

SUMMARY:
Open heart surgery, including coronary artery bypass grafting (CABG) and/or aortic valve replacement (AVR) is associated with a significant risk of mortality.

This study is a randomized clinical trial with the purpose of investigating four different interventions on the primary endpoint 'days alive and outside of hospital within 90 days'.

The interventions are:

* Dexamethasone vs. placebo administered after induction of anesthesia.
* Olanzapine vs. placebo administered prior to anesthesia.
* A blood-flow targeted vs. a blod-pressure targeted hemodynamic strategy while the patient is on cardio-pulmonary bypass (CPB)
* Low-tidal volume ventilation vs. no ventilation of the lungs while the patient is on CPB

DETAILED DESCRIPTION:
1. BACKGROUND

   1.1 Coronary artery bypass grafting and valve replacement Open heart surgery, including coronary artery bypass grafting (CABG) and/or aortic valve replacement (AVR) is associated with a significant risk of mortality. Elective CABG remains associated with a mortality of approximately 1.5 % after 30 days and increases to approximately 9 % after 5 years, with higher percentages in the subacute setting. Aortic valve replacement (AVR) is associated with a mortality of approximately 6% after 30 days, while mitral valve replacement (MVR) is associated with a mortality of approximately 4%. Additionally, open heart surgery is associated with a significant risk of morbidity caused by organ injury, including multi-organ failure, cerebral injury, pulmonary injury, cardiac injury, renal injury and/or endothelial injury.

   1.2 Organ injury associated with cardiac surgery and cardiopulmonary bypass The primary indication for CABG with/without AVR is atherosclerotic disease with associated coronary artery disease and/or valvular disease. Atherosclerotic disease may affect the perfusion and function of other organs, such as the brain, heart, lungs and kidneys, and make them vulnerable to the homeostatic changes that occur during open heart surgery. As such, pre-existing organ disease increases the risk of organ injury, and the clinically applied risk scores 'European System for Cardiac Operative Risk Evaluation' (EuroSCORE II) and 'Society of Thoracic Surgeons' (STS) score both include extracardiac vascular disease, heart failure, kidney function and lung disease, as independent predictors of in-hospital or 30-day mortality after open heart surgery. During CABG/AVR, extracorporeal circulation is applied in the form of cardiopulmonary bypass (CPB). Changes in blood flow occur during initiation and weening of CPB and also as a consequence of the fixed, non-pulsatile flow of the CPB circuit. These flow changes may affect end-organ perfusion, cause reperfusion injury, trigger inflammatory cascades and play a part in ensuing morbidity or mortality. Furthermore, open heart surgery induces severe systemic inflammation caused by the surgical procedure itself (sternotomy and ensuing lung collapse) as well as the result of mechanical stress and exposure to the artificial surfaces of the CPB circuit for the blood.

   1.3 Dexamethasone The use of glucocorticoids for mitigation of the inflammatory response during cardiac surgery has been investigated previously. In earlier studies, the use of prophylactic glucocorticoids have been suggested to lower the risk of post-operative atrial fibrillation, reduce post-operative bleeding, shorten the duration of mechanical ventilation and the length of stay in the intensive care unit (ICU) as well as shorten length of hospital stay. However, these earlier clinical trials have been assessed mostly as being of low quality and underpowered to draw conclusions regarding patient-centred outcomes. In non-cardiac surgery, the use of low to intermediate dose glucocorticoids have been suggested to have opioid-sparing effects and to decrease post-operative pain as well as nausea and vomiting.

   Two large, well-conducted randomized clinical trials (RCTs) have investigated high-dose glucocorticoid prophylaxis in patients undergoing CPB. In the Dexamethasone for Cardiac Surgery (DECS) trial, a total of 4,494 patients undergoing heart surgery with CPB were randomized to a single intraoperative dose of 1mg/kg of dexamethasone versus placebo. The study found no significant difference in a composite endpoint consisting of death, myocardial infarction (MI), stroke, renal failure or respiratory failure within 30 days of randomization (relative risk (RR) 0.83 (95%CI 0.67 - 1.01, p=0.07). Dexamethasone was associated with a reduction in postoperative infection, the need for mechanical ventilation and reduced length of ICU and hospital stay and with higher postoperative glucose levels. In the Steroids In cardiac Surgery (SIRS) trial, a total of 7,507 patients undergoing cardiac surgery with CPB were randomized to a total of 500mg of methylprednisolone versus placebo, initiated in the operating room. The study found no significant difference in 30-day mortality between the groups (RR 0.87 (95%CI 0.70 - 1.07, p=0.19). Furthermore, the study found no significant differences in the pre-specified safety outcomes with the exception of higher blood glucose levels in the patients who received methylprednisolone. A patient-level meta-analysis of the DECS SIRS trials show a reduction in the rates of respiratory failure and infections in favour of glucocorticoids while glucocorticoids were associated with an increase in myocardial injury but not MI as defined by the 3rd universal definition. Both the DECS and the SIRS trial used high dose glucocorticoids. A previous dose-response meta-analyses have suggested that low dose glucocorticoids maybe beneficial compared to high dose glucocorticoids. Accordingly, for non-cardiac surgery, lower doses of glucocorticoids of between 0.1 mg/kg to 0.2 mg/kg are frequently applied, which may balance positive effects with adverse effects.

   1.4 Olanzapine Delirium and post-operative cognitive dysfunction are frequent following cardiac surgery. The risk of delirium is approximately 30% and it has been associated with a decline in activities of daily living after 6 months. Cognitive decline after non-cardiac surgery has been associated with increased mortality. Olanzapine is a second-generation antipsychotic that have exhibited affinity to a range of receptors, including serotonin, dopamine, cholinergic, and histamine receptors in preclinical studies. The main indications of olanzapine include treatment of schizophrenia and moderate-to-severe manic episode. For treatment of delirium in the ICU, olanzapine has been suggested as an alternative to haloperidol, exhibiting less extrapyramidal side effects. Several studies have shown that olanzapine are associated with minimal changes in the electrocardiogram QT interval. In 2010, Larsen et al. showed that 5mg of olanzapine administered prior to surgery as well as immediately after surgery reduced delirium in 495 patients undergoing joint replacement (knee or hip). The incidence of postoperative delirium from surgery to discharge was 14% in the olanzapine group versus 40% in the placebo group (p < 0.0001). Later meta-analyses and reviews conclude that there is insufficient data to draw conclusions regarding the effects of antipsychotics for postoperative delirium prophylaxis, but suggest that olanzapine is among the promising drugs.

   1.5 Hemodynamic management during cardiopulmonary bypass While the pathophysiology behind organ injury in relation to CPB is complex, the balance between oxygen delivery (DO2) and oxygen consumption (VO2) to the organs is likely to play an important role in organ injury. The DO2 can be approximated as a product of pump flow, haematocrit (HCT), and arterial oxygen saturation (SaO2), while the VO2 can be approximated as the difference between SaO2 and central venous oxygen saturation (ScvO2). Previously, a low DO2 during CPB has been associated with postoperative delirium and kidney injury. In contrast, a recent multicentre RCT found that maintaining a DO2 target above 280mL per minute per square meter body surface area reduced the incidence of acute kidney injury stage I in 350 patients undergoing CPB. Contemporary guidelines on CBP in adult cardiac surgery suggest that the adequacy of the pump-flow rate should be checked based on oxygenation parameters, and that the pump-flow should be adjusted according to arterial oxygen content (i.e. haematocrit and SaO2). However, equipoise exists regarding the specific DO2 targets, and how to increase DO2.

   Targeting a sufficient mean arterial pressure (MAP) is likely important to ensure an adequate perfusion pressure to the organs. The perfusion pressure can be approximated as the difference between MAP and central venous pressure. During CPB, the MAP can be targeted either by regulation of pump flow or by administration of vasopressors. Increased CPB flow rate has been proposed to be associated with increased haemolysis, hypertension during hypothermic CPB, and increased risk of embolization (from a theoretical standpoint). Previously, 4 RCTs have compared a higher to a lower MAP strategy. The largest trial by Charlson et al randomized 412 patients to a target MAP of 80 mmHg versus a custom MAP defined by pre-CPB pressure, and found no significant difference in outcomes between groups. In contrast, Siepe et al reported less delirium and early cognitive dysfunction in 44 patients randomized to a high MAP target of 80-90 mmHg compared to 48 patients randomized to a low MAP target of 60-70 mmHg. Gold et al randomized 124 patient to either a MAP of 80-100 mmHg or a MAP of 50-60 mmHg, and found a difference in favour of the high MAP target for a composite endpoint of neurologic and cardiac morbidity. Most recently, Vedel et al randomized 197 patients to a high MAP target of 70-80 mmHg versus a low MAP target of 40-50 mmHg and found no differences in postoperative cerebral infarcts assessed by magnetic resonance diffusion weighted imaging, postoperative cognitive dysfunction, levels of biomarkers reflecting cerebral injury or long-term survival or cognitive function. Accordingly, equipoise exists regarding the optimal MAP during CPB and contemporary guidelines recommend a relative wide MAP interval from 50 to 80 mmHg during CPB.

   1.6 Ventilation and positive end-expiratory pressure (PEEP) during cardiopulmonary bypass (CPB) Postoperative pulmonary complications are common after on-pump cardiac surgery, ranging from mild hypoxemia to acute respiratory distress syndrome. Pulmonary complications are associated with risk of re-intubation and prolonged ICU stay and have been attributed to approximately 26% of in-hospital mortality after cardiac surgery. Maintaining mechanical ventilation or a positive airway pressure during CPB has been shown to improve gas exchange post-operatively, and higher PEEP have been shown to reduce atelectasis and inflammation in cardiac surgery. Two recent studies, the PROVECS trial and the MECANO trial, have examined open-lung versus conventional perioperative ventilation strategies during CPB in cardiac surgery. In the PROVECS trial, 493 patients were randomized 1:1. Patients in the intervention group were randomized to low volume ventilation (TV 3ml/kg, PEEP 8 cm H20, FiO2 0.4) with intermittent recruitment manoeuvres at PEEP 30cm H20 for 30 seconds. The control group was randomized to a set PEEP of 2 cm H2O. Postoperative pulmonary complications (a composite primary endpoint) occurred in 55% of patients in the intervention group and in 59% in the control group (p=0.32). In the MECANO trial, 1,501 patients were randomized. Patients in the intervention group received low volume ventilation (TV 3ml/kg, PEEP 5 cm H20), while the control group received no ventilation and no PEEP. The composite outcome of death, early respiratory failure, ventilatory support after day 2 and reintubation occurred in 15% in the ventilation group versus 18% in the no-ventilation group (Odds ratio (OR) 0.80 (0.61-1.05, p=0.11)). In patients undergoing isolated CABG, the ventilation strategy was superior for the primary outcome (OR 0.56 (0.37-0.84, p=0.005)). Accordingly, equipoise exists for the ventilation strategy during CPB, which is supported by contemporary reviews and meta-analyses. Contemporary guidelines suggest that PEEP during CBP should be considered and that ventilation during CPB may be considered for lung protection. The methodological quality of the RCTs in the meta-analysis informing the guidelines recommendation was graded as low.
2. TRIAL OBJECTIVES

2.1 Primary objective The primary objective of this trial is to determine the efficacy of dexamethasone compared with placebo on the primary endpoint days alive outside hospital within 90 days in adult subjects undergoing elective or subacute isolated CABG, isolated AVR, or CABG plus any concomitant valve surgery. The coprimary objectives are to determine the efficacy of olanzapine versus placebo administered preoperatively, the efficacy of flow-targeted versus pressure-targeted hemodynamic management during CPB, and the efficacy of low tidal volume ventilation versus no ventilation during CPB, on the endpoint days alive outside hospital within 90 days in adult subjects undergoing elective or subacute isolated CABG, isolated AVR, or CABG plus any concomitant valve surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, i.e., above 18 years of age
2. Scheduled for CABG and/or AVR, irrespective of other concomitant valve surgery.

Exclusion Criteria:

1. Acute surgery (i.e. off hours surgery)
2. Pregnancy or currently breastfeeding. Pregnancy in all fertile women will be ruled out by pregnancy testing prior to randomization.
3. Known endocarditis at time of screening
4. Previous participation in the trial
5. Active infection, including bacterial, viral, and/or fungal infection
6. Known hepatic cirrhosis
7. Known severe thrombocytopenia with thrombocyte levels < 50 x 109/L
8. Known severe neutropenia with neutrocyte levels < 2 x 109/L
9. On the waiting list for a heart transplant
10. Recipient of any major organ transplant
11. Obstructive hypertrophic cardiomyopathy, active myocarditis, constrictive pericarditis, untreated hypothyroidism or hyperthyroidism
12. Having received cytotoxic/cytostatic chemotherapy or radiation therapy for treatment of malignancy within the last 6 months.
13. Clinical evidence of current malignancy except for basal or localized squamous cell carcinoma, cervical intraepithelial neoplasia or stable prostate cancer.
14. Known narrow-angle glaucoma
15. Known phenylketonuria
16. Type I diabetes
17. Known long QT syndrome
18. Known allergy for any of the included study drugs
19. Any condition, where participation in the study, in the investigator's opinion could put the subject at risk, confound the study results or interfere significantly with participation in the study

Patients with extracardiac arteriopathy (assessed as part of the pre-operative EuroSCORE) will be excluded from the intervention 'flow-targeted vs. pressure-targeted hemodynamic management during CPB'.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Days alive and outside hospital | 90 days from surgery

SECONDARY OUTCOMES:
Time to composite outcome of death and major organ damage | 90 days
  Time in days to occurrence of any component in a composite secondary endpoint during follow-up consisting of
  1. Death from any cause
  2. Stroke, defined as persisting (>24 hours) of any neurological symptoms of neurological dysfunction during the 6 months follow-up period. The diagnosis is determined by the treating physician.
  3. Acute kidney injury requiring any type of renal replacement therapy during the follow-up period.
  4. New onset or worsening heart failure, defined as persistent (> 24 hours from initiation) need for vasopressor/inotropic hemodynamic support, need for mechanical circulatory support after surgery, inability to close the sternotomy due to hemodynamic instability after surgery or readmission for acute heart failure during follow-up.
Number (fraction) of patients with severe post-operative complications during index admission, defined as a Clavien-Dindo class of 3 to 5. | During index admission up to 30 days after surgery. Outcome will be assessed upon hospital discharge.
  The Clavien-Dindo classification runs from 1 to 5 with a higher score indicating more severe complications.
Number (fraction) of patients with delirium, defined as a positive Confusion Assessment Method for the ICU (CAM-ICU) or wards (CAM). | During index admission up to 30 days after surgery.
  Number (fraction) of patients with delirium during index admission will be reported. Outcome will be assessed daily until hospital discharge.
Quality of Recovery-15 (QoR-15) score | 3 days or as soon as possible after surgery
  The QoR-15 score includes 15 questions with each question being graded from 0-10.
Survival | Within 90 days
Graft patency, assessed by cardiac computed tomography (CT) scan | After 90 days
Myocardial resting perfusion, assessed by cardiac CT scan | After 90 days
Change in modified Rankin Scale (mRS) from baseline | After 90 days
  Score ranging from 0 to 6, with a higher score indicating a worse outcome.
Health-related quality of life (EQ-5D-5L) | After 90 days
  5 dimensions and 5 questions with higher scores indicating a worse outcome.
Change in self-perceived function "two simple questions" | After 90 days
  Two questions: 'Have you within the past two weeks needed help for every day activities', and 'Do you feel that you have recovered completely after your operation'
Days alive outside ICU within 90 days | 90 days
Survival | 180 days

OTHER OUTCOMES:
Surgical wound infection | Within 90 days
  Surgical wound infection including sternum infection and/or endocarditis, requiring antibiotics for > 48 hours and/or surgical revision.
Sepsis | Within 90 days
  Sepsis, as defined by the Sepsis-3 criteria, requiring antibiotics for a minimum of 3 consecutive days.
  3)
Acute kidney injury | Within 90 days
  Acute kidney injury, as defined by the KDIGO criteria.
Myocardial infarction | Within 90 days
  Myocardial infarction, as defined by the Fourth Universal Definition of Myocardial Infarction.
Bleeding | Within 90 days
  Post-surgical bleeding requiring transfusion
Readmission | Within 90 days
Re-operation for any cause | Within 90 days
  This endpoint will be stratified by major causes.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hassager, MD, DMSc, Study Chair — Sponsor GmbH
Locations (1):
- The Heart Centre, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No